CLINICAL TRIAL: NCT06258681
Title: Examining the Clinical Efficiency of a Customizable Respiratory Exercise Device in Individuals Who Have Undergone Cardiac Surgery
Brief Title: Customizable Respiratory Exercise Device in Individuals Who Have Undergone Cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Collaborators: Istanbul Galata University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, Assoc. Prof., Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 682201
Record Dates: First submitted 2024-01-26; First posted 2024-02-14 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease
Keywords: cardiac surgery; respiratory muscle training; aerobic exercise
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: This is a two-arm controlled single blind trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: The assessor will be blind to the group allocation and participants will be blind to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Incentive spirometry group (Active Comparator): The incentive spirometry group will continue the 8-week training with Volumetric Triflo. Individuals will be expected to exhale normally and hold their breath for at least 3 seconds after taking as deep a breath as possible. In the first week after surgery, the individual will be asked to work with an incentive spirometry in 10 repetitions every hour when awake. The group also followed standard program which includes phases of chest physiotherapy (modified postural drainage and assisted coughing techniques) and early progressive mobilization (gradually increasing walking distance in the corridor depending on patient tolerance). Participants in both groups will continue aerobic exercise training in the clinic until the end of the 8th week after discharge. Aerobic exercise training includes a bicycle ergometer, two days a week, 20-30 minutes, and perceived effort in the range of 60-70% of the maximal heart rate, in the range of 4-6 according to the Modified Borg Scale.
  Interventions: Other: Incentive spirometer
- Individualized respiratory training group (Experimental): In the first week after surgery, the personalized breathing exercise device will be adjusted to the resistance level corresponding to 40% of the initial pressure load, MIP, and MEP measurements. Participants will be asked to rest and repeat the training for ten sets following five breathing cycles. In each set, there will be a one-minute rest break between repetitions. Participants can practice both inspiratory and expiratory respiratory muscle training in a single breathing cycle. As the progression progresses, the perceived exertion level will be increased by 5-10% every week to a range of 4-6 according to the Modified Borg Scale. The training will continue for eight weeks.
  Interventions: Other: Individualized respiratory training group

INTERVENTIONS:
Other: Incentive spirometer — The incentive spirometry group will continue training with Volumetric Triflo. It is asked to exhale at first and then hold their breath for at least 3 seconds after taking as deep a breath as possible.
  Arms: Incentive spirometry group
Other: Individualized respiratory training group — Participants will be able to practice both inspiratory and expiratory respiratory muscle training in a single breathing cycle.
  Arms: Individualized respiratory training group

SUMMARY:
The cardiorespiratory system integrates systemic and pulmonary circulation while ensuring adequate oxygenation of the body at rest and during exercise. In addition to chronic respiratory problems that mainly affect the lungs, airways and pulmonary vascular system, respiratory capacity and respiratory muscle strength can be negatively affected in a wide spectrum including cardiac diseases, surgeries, neuromuscular diseases, obesity, long-term bed rest, aging and inactivity. Weakness of the respiratory muscles causes important secondary consequences by causing the increased respiratory demands not to be met during physical activity. It has been reported that respiratory muscle training applied within the scope of pre-operative and post-operative cardiac rehabilitation program is beneficial in terms of increasing respiratory functions, reducing the risk of post-operative complications and length of stay. Respiratory muscle training is known to have many potential beneficial effects on patients undergoing cardiac surgery. Different methods and devices are used to improve and develop the functions of the inspiratory and expiratory muscles and each training method and device has differences. Therefore, it is thought that examining the clinical effects of using a personalized breathing exercise device on respiratory functions, respiratory muscle strength and functional capacity in individuals who have undergone cardiac surgery will contribute to the literature.

DETAILED DESCRIPTION:
Breathing exercises can be applied specifically to different segments of the lungs, increasing collateral ventilation and helping mobilize secretions. Chronic respiratory diseases, rib cage deformities, neuromuscular diseases that cause breathing problems, lung transplant or lung surgery patients in the pre-operative and post-operative period, cancer patients, heart failure patients and cardiovascular surgery patients, and those whose quality of life is impaired due to shortness of breath. People are known to be groups that benefit from breathing exercises. Breathing exercises have been shown to be effective in preserving respiratory function and preventing or reducing respiratory complications in all of these conditions. It has been reported that respiratory muscle training applied within the scope of pre- and post-operative cardiac rehabilitation programs is beneficial in increasing respiratory functions and reducing the risk of postoperative complications and length of stay. Respiratory muscle training is known to have many potential beneficial effects on patients undergoing cardiac surgery. Different methods and devices are used to improve and develop the functions of inspiratory and expiratory muscles, and each training method and device has differences. For this reason, the respiratory exercise device to be developed is aimed to be a device that can be shaped according to the desired purpose, has visual feedback, and can combine multiple respiratory muscle training methods. The device is thought to play an active role in rehabilitating complications such as lung ventilation and respiratory muscle weakness, which are frequently affected in patients after major surgery such as cardiac surgery. Therefore, it is thought that examining the clinical effects of using a personalized breathing exercise device on respiratory functions, respiratory muscle strength, and functional capacity in individuals who have undergone cardiac surgery will contribute to the literature.

ELIGIBILITY:
Inclusion criteria

* Individuals with New York Heart Association Functional Class I or II who are scheduled to undergo elective coronary artery bypass graft surgery, aortic valve replacement, mitral valve replacement, or combined surgery of aortic and mitral valve replacement
* Individuals who are planning to undergo surgery with the median sternotomy technique
* Individuals with Mini-Mental State Score >24

Exclusion criteria

* Individuals with uncontrolled arrhythmia, unstable angina pectoris, uncontrolled hypertension
* Individuals with accompanying chronic respiratory disease
* Individuals with accompanying neuromuscular or orthopedic/musculoskeletal limitations
* Individuals with a history of spontaneous or trauma-related pneumothorax
* Individuals with middle ear-related pathologies (such as tympanic membrane rupture otitis)
* Cases with thorax drains in the ward
* Individuals who stayed in the intensive care unit for ≥ 4 days in the postoperative period
* Individuals who have had another surgery in the last six months

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
The Forced Expiratory Volume 1st second | 8 weeks
  The volume of air exhaled in the 1st second of forced expiration will be noted.
Forced Vital Capacity | 8 weeks
  The volume of air exhaled rapidly and forcefully following deep inspiration will be noted.
Peak Expiratory Flow | 8 weeks
  Maximum inspiration followed by maximum exhalation maneuver will be measured and noted.
Respiratory Muscle Strength | 8 weeks
  Inspiratory and expiratory respiratory muscle strength will be evaluated by intraoral pressure measurement method.
Six minutes walking test | 8 weeks
  Functional capacity evaluation will be done with 6 Minute Walking Test. Six minutes walking distance will be noted.

SECONDARY OUTCOMES:
Minnesota Life with Heart Failure Questionnaire. | 8 weeks
  Quality of life will be assessed using the Minnesota Life with Heart Failure Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Ezelsoy, MSc, Study Director — Bilim University
Locations (1):
- Istanbul Florence Nightingale Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No